CLINICAL TRIAL: NCT00623103
Title: A 76-week Prospective, Open-label, Multicenter Study to Evaluate the Long-term Effect of Rivastigmine Capsule and Transdermal Patch on Worsening of the Underlying Motor Symptoms of PD in Patients With Mild to Moderately Severe Dementia Associated With Parkinson's Disease (PDD)
Brief Title: Long-term Safety of Rivastigmine Capsule and Patch in Patients With Mild to Moderately-severe Dementia Associated With Parkinson's Disease (PDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CENA713B2315
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-10

CONDITIONS: Parkinson's Disease Dementia
Keywords: Parkinson's disease dementia; cholinesterase inhibitor; rivastigmine
MeSH Terms: interventions — Rivastigmine

ARMS (2):
- Rivastigmine capsule (Experimental): Rivastigmine capsules starting at a total dose of 3 mg/day (1.5 mg twice daily orally) titrated up in 3 mg/day increments every 4 weeks to a final dose of 12 mg/day (6 mg twice daily orally). The 12 mg/day dose or the highest dose tolerated was maintained until week 76.
  Interventions: Drug: Rivastigmine capsule
- Rivastigmine patch (Experimental): Rivastigmine patch once a day in the morning, worn for 24 hours, starting at 5 cm^2 (delivering 4.6 mg rivastigmine over a 24 hour period) for 4 weeks then titrated up to 10 cm^2 daily (delivering 9.5 mg rivastigmine over a 24 hour period). The 10 cm^2 patch or the highest well tolerated dose was maintained until week 76.
  Interventions: Drug: Rivastigmine transdermal patch

INTERVENTIONS:
Drug: Rivastigmine capsule — Rivastigmine capsules orally twice a day. Target dose 12 mg/day.
  Other Names: Exelon®
  Arms: Rivastigmine capsule
Drug: Rivastigmine transdermal patch — Rivastigmine patch once a day in the morning, worn for 24 hours. Target dose 10 cm^2/day delivering 9.5 mg over a 24 hour period.
  Other Names: Exelon®
  Arms: Rivastigmine patch

SUMMARY:
The purpose of this study is to provide long-term safety data for rivastigmine capsule and transdermal patch treatments, in particular the effect of rivastigmine on worsening of the underlying motor symptoms of Parkinson's Disease (PD), in patients with mild to moderately severe dementia associated with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease, according to the UK Parkinson's disease Society Brain Bank criteria
* Diagnosis of Parkinson's disease dementia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria, with onset of symptoms of dementia at least 2 years following the first diagnosis of idiopathic Parkinson's disease
* Mini Mental State Examination score of ≥10 and ≤ 26 (at Screening Visit only)

Exclusion Criteria:

* An advanced, severe, or unstable disease of any type that may interfere with the primary and secondary variable evaluations
* A score of 5 (wheelchair bound or bedridden) in the "on"-state on the Modified Hoehn and Yahr Staging (UPDRS Part V)
* A current diagnosis of any primary neurodegenerative disorder other than idiopathic PD
* A current diagnosis of any treatable dementia (hypothyroidism, syphilis, vitamin B12 or folate deficiency) that is verified by the investigator to be the cause of dementia.
* A current diagnosis of probably vascular dementia according to the National Institute of Neurological Disorders and Stroke and the Association International pour la Recherche et l'Enseignement en Neurosciences (NINDS-AIREN) criteria
* A current diagnosis of a major depressive episode according to DSM-IV criteria
* A history of stereotaxic brain surgery for Parkinson's disease
* A known exaggerated pharmacological sensitivity or hypersensitivity to drugs similar to rivastigmine or to other cholinergic compounds

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (118):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - 21st Century Neurology, Phoenix, Arizona
  - Neurosearch, Inc., Reseda, California
  - Neurosearch II, Inc., Ventura, California
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Comprehensive Neurology Specialists, PC, Suwanee, Georgia
  - Neurological Associates, Meridian, Idaho
  - Evanstan Northwestern Healthcare Medical Group, Glenview, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Neurological Care of Central NY, Syracuse, New York
  - Neurology & Neuroscience Associates, Inc., Akron, Ohio
  - Square 1 Clinical Research, Erie, Pennsylvania
  - Research Protocol Management Solutions, Pittsburgh, Pennsylvania
  - Neurology Specialists of Dallas, Dallas, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Veterans Affairs Puget Sound Health Care System, Seattle, Washington
- Argentina (4):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Buenos Aires F.D.
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Australia (5):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Malvern, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Prahran, Victoria
- Austria (5):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (8):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Wilrijk
- Canada (12):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
- France (9):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Clermont
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative site, Pessac
  - Novartis Investigative site, Rennes
  - Novartis Investigative Site, Roanne
- Germany (19):
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Beelitz-Heilstätten
  - Novartis Investigative site, Berlin
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Leun-Biskirchen
  - Novartis Investigative Site, Lubin
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative site, Ulm
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wolfach
- Italy (12):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Lido di Camaiore, LU
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Arcugnano, VI
  - Novartis Investigative site, Cassino
  - Novartis Investigative Site, Napoli
- Netherlands (10):
  - Novartis Investigative Site, Zwolle, AB
  - Novartis Investigative Site, Blaricum, AN
  - Novartis Investigative Site, Maastricht, AZ
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, Enschede, ER
  - Novartis Investigative Site, Tilburg, GC
  - Novartis Investigative Site, Groningen, GZ
  - Novartis Investigative Site, 's-Hertogenbosch, JL
  - Novartis Investigative Site, Heerlen, PC
  - Novartis Investigative Site, Sittard
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Sihhiye/Ankara
  - Novartis Investigative Site, Yenisehir/Izmir
- United Kingdom (8):
  - Novartis Investigative Site, Blackburn
  - Novartis Investigative Site, Blandford Forum, Dorset
  - Novartis Investigative Site, Christchurch, Dorset
  - Novartis Investigative Site, Newcastle
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Peterborough
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Vale of Glamorgan

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivastigmine Capsule: Rivastigmine capsules starting at a total dose of 3 mg/day (1.5 mg twice daily orally) titrated up in 3 mg/day increments every 4 weeks to a final dose of 12 mg/day (6 mg twice daily orally0. The 12 mg/day dose or the highest dose tolerated was maintained until week 76.
Period: Overall Study
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Started | 295 | 288
Safety Set: Received Study Drug | 294 (One randomized participant did not receive study drug and was not included in the Safety set.) | 288
Completed | 184 | 175
Not Completed | 111 | 113
Not completed — Adverse Event | 70 | 60
Not completed — Unsatisfactory therapeutic effect | 4 | 12
Not completed — Withdrawal by Subject | 18 | 24
Not completed — Lost to Follow-up | 4 | 1
Not completed — Administrative problems | 2 | 4
Not completed — Death | 11 | 11
Not completed — Protocol deviation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch | Total
Number analyzed (Participants) | 295 | 288 | 583
Age Continuous [Mean (Standard Deviation); unit: years] | 72.35 (6.295) | 72.26 (6.352) | 72.31 (6.318)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 97 | 185
  Male | 207 | 191 | 398

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Due, or Potentially Due, to Worsening of Parkinson Disease (PD) Motor Symptoms (Tremor, Muscle Rigidity, Bradykinesia, Fall)
Description: The AEs were summarized by presenting the number and percentage of patients having any of the 4 AEs or discontinued due to any of the 4 predefined AEs (tremor, muscle rigidity, bradykinesia, and fall)in each treatment group. The 95% CIs associated with the rates were also presented.
Time Frame: 76 Weeks
Population: Safety Population consisted of all participants who received at least 1 dose of study drug and had 1 post-baseline safety measurement. Participants with observation at 76 weeks were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Number analyzed (Participants) | 294 | 288
Percentage of participants
  Tremor | 24.5 [19.7 to 29.8] | 9.7 [6.6 to 13.7]
  Muscle Rigidity | 4.1 [2.1 to 7.0] | 5.2 [2.9 to 8.4]
  Bradykinesia | 5.1 [2.9 to 8.3] | 6.3 [3.7 to 9.7]
  Fall | 17.0 [12.9 to 21.8] | 20.1 [15.7 to 25.2]

2. Primary Outcome: Percentage of Participants With Study Drug Discontinuations Due to Predefined AEs That Are Due, or Potentially Due, to Worsening of PD Motor Symptoms (Tremor, Muscle Rigidity, Bradykinesia, Fall)
Description: The discontinuations due to these AEs were summarized by presenting the number and percentage of patients having any of the 4 AEs or discontinued due to any of the 4 predefined AEs (tremor, muscle rigidity, bradykinesia, and fall) in each treatment group. The 95% CIs associated with these rates were also presented.
Time Frame: 76 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Number analyzed (Participants) | 294 | 288
Percentage of participants
  Tremor | 2.4 [1.0 to 4.8] | 0.7 [0.1 to 2.5]
  Muscle Rigidity | 0.3 [0.0 to 1.9] | 0.3 [0.0 to 1.9]
  Bradykinesia | 1.0 [0.2 to 3.0] | 0.0 [0.0 to 0.0]
  Fall | 1.0 [0.2 to 3.0] | 1.4 [0.4 to 3.5]

3. Secondary Outcome: Change in Unified Parkinson Disease Rating Scale (UPDRS) Part III Motor Examination Scores at Weeks 8, 16, 24, 52 and 76 (or Early Discontinuation) Compared to Baseline
Description: Unified Parkinson Disease Rating Scale (UPDRS) is a 6 part Parkinson's disease specific rating scale that estimates clinical function taking into consideration both disability (functional deficits) and impairment (objective clinical signs). Part III records the motor examination in Items 18-31 rated on a scale of 0 to 4 with (0 being absent/ normal and 4 being the worse) for a total possible score of 0 to 56.
Time Frame: From Baseline to Weeks 8, 16, 24, 52 and 76
Population: Safety population consisted of all participants who received at least 1 dose of study drug and had 1 post-baseline safety measurement. "n" in each of the categories is the number of participants at each time point with non-missing baseline and post-baseline measurements.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Number analyzed (Participants) | 294 | 288
Score on a scale
  Week 8 (n=276,277) | -0.4 (6.99) | -0.9 (7.05)
  Week 16 (n=254,252) | 0.5 (7.72) | -1.7 (7.44)
  Week 24 (n=229,237) | 0.1 (8.19) | -1.4 (7.90)
  Week 52 (n=203,206) | 0.7 (8.66) | 1.6 (9.57)
  Week 76 (n=183,175) | 2.1 (9.98) | 2.1 (9.65)

4. Secondary Outcome: Change in Mattis Dementia Rating Scale (Mattis DRS-2) Scores at Weeks 16, 24, 52 and 76 Compared to Baseline
Description: Mattis DRS-2 is a measure of cognitive status. The total score is the sum of 5 subscale scores: Attention [0-37], Initiation/Perservation [0-37] (performing alternating movements), Construction [0-6] (copying designs), Conceptualization [0-39] (similarities) and Memory [0-25] (sentence recall, design recognition)for a total possible score of 0-144. Higher score is reflective of better cognitive function, lower scores associated with more pronounced cognitive deficit. The change from baseline was calculated such that a positive number indicates an improvement.
Time Frame: From Baseline to Weeks 16, 24, 52 and 76
Population: Intent-to-treat population which included all patients who received at least 1 dose of study drug and had at least 1 pre- and post-baseline assessment for 1 of the efficacy variables. Last observation carried forward. (LOCF)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Number analyzed (Participants) | 273 | 273
Score on a scale
  Week 16 | 5.4 (11.98) | 3.4 (11.53)
  Week 24 | 6.5 (12.98) | 4.4 (12.85)
  Week 52 | 4.6 (13.62) | 1.3 (15.07)
  Week 76 | 3.9 (16.82) | -1.4 (17.43)

5. Secondary Outcome: Change in Ten Point Clock Test (TPCT) Scores at Weeks 16, 24, 52 and 76 (or Early Discontinuation) Compared to Baseline
Description: The Ten Point Clock Test measures executive functioning and visuospatial skills. Participants are asked to put numbers on the face of a clock and then make the clock read 10 minutes after 11. Points are awarded on a scale of 0 to 10 for spacing of specific numbers and the positions of the hands. The change from baseline was calculated such that a positive number indicates improvement.
Time Frame: From Baseline to Weeks 16, 24, 52 and 76
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Number analyzed (Participants) | 273 | 273
Score on a scale
  Week 16 | 0.5 (2.75) | 0.4 (3.02)
  Week 24 | 0.6 (3.18) | 0.3 (3.40)
  Week 52 | 0.3 (2.97) | -0.1 (3.33)
  Week 76 | 0.0 (3.2) | -0.3 (3.57)

6. Secondary Outcome: Change in Neuropsychiatric Inventory-10 (NPI-10) Scores at Weeks 16, 24, 52 and 76 (or Early Discontinuation) Compared to Baseline
Description: The parameter for analysis was the change from baseline of total score of 10 items on the NPI scale (NPI-10). The total score is a sum of the 10 domains, where the score for a domain is defined as the product of frequency (range: 1-4) and severity (range: 1-3). Each domain has a maximum score of 12 and all domains were equally weighted for total score(thus the range for the total score is 0 to 120 with 0 being completely healthy to 120 which is the worse score patient can get). The change from baseline was calculated such that a negative number indicates an improvement (symptom reduction).
Time Frame: At Week 16, 24, 52 and 76 (or early discontinuation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Number analyzed (Participants) | 294 | 288
Score
  Week 16 | -3.3 (9.75) | -0.5 (10.89)
  Week 24 | -2.6 (10.31) | -1.0 (10.27)
  Week 52 | -1.7 (11.40) | -0.3 (11.26)
  Week 76 | -1.6 (11.22) | 0.7 (12.62)

7. Secondary Outcome: Change in Alzheimer's Disease Cooperative Study-Activities Of Daily Living (ADCS-ADL) Scores at Weeks 16, 24, 52 and 76 (or Early Discontinuation) Compared to Baseline
Description: The 23 item caregiver-based ADL scale of the dementia Alzheimer's disease Cooperative Study-Activities of Daily Living (ADCS-ADL) was used for analysis. This is a caregiver rated questionnaire of 23 items, with possible scores over a range of 0-78, where 78 denote full functioning with no impairment. The total score was derived by adding up the item scores of the 23 items.
  The change from baseline was calculated such that a positive change indicates an improvement.
Time Frame: From Baseline to Week 16, 24, 52 and 76 (or early discontinuation)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Number analyzed (Participants) | 294 | 288
Score
  Week 16 (n=273, 270) | -0.4 (9.60) | -1.3 (10.38)
  Week 24 (n=273,270) | -0.6 (10.12) | -1.5 (10.91)
  Week 52 (n=273,270) | -2.2 (11.13) | -5.4 (13.57)
  Week 76 (n=273, 270) | -4.4 (13.13) | -7.8 (15.62)

8. Secondary Outcome: UPDRS Part V Stage (Modified Hoehn and Yahr Staging)at Baseline, Week 8,16,24,52 and 76 (or Early Discontinuation)
Description: Unified Parkinson Disease Rating Scale (UPDRS) is a 6 part Parkinson's disease specific rating scale that estimates clinical function taking into consideration both disability (functional deficits) and impairment (objective clinical signs). UPDRS Part V is assessed by the modified Hoehn and Yahr Staging Scale. The scale ranges from 0 (no signs of disease) to 5 (wheelchair bound or bedridden unless aided).
Time Frame: From Baseline to Week 8, 16, 24, 52 and 76 (or early discontinuation)
Population: The Safety population consisted of all patients who have received at least one dose of study drug and have had at least 1 safety measurement after baseline. n=indicates patients with observation during different timepoints.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Rivastigmine Capsule | Rivastigmine Patch
Number analyzed (Participants) | 294 | 288
Score
  Baseline (n = 294,288) | 2.7 (0.65) | 2.7 (0.70)
  Week 8 (n=17,18) | 2.6 (0.70) | 2.7 (1.05)
  Week 16 (n=254,252) | 2.8 (0.68) | 2.7 (0.67)
  Week 24 (229, 236) | 2.7 (0.75) | 2.7 (0.67)
  Week 52 (n=202,208) | 2.8 (0.73) | 2.8 (0.69)
  Week 76 (n=184, 175) | 2.8 (0.74) | 2.8 (0.79)

ADVERSE EVENTS:
Groups:
- Exelon Capsule: Exelon Capsule
- Exelon Patch: Exelon Patch
Arm/Group | Exelon Capsule | Exelon Patch
Serious Adverse Events (participants affected / at risk) | 87/294 | 83/288
Other Adverse Events (participants affected / at risk) | 239/294 | 215/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exelon Capsule (N=294) | Exelon Patch (N=288)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac valve sclerosis (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mesenteric occlusion (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Complication of device insertion (General disorders) | 0 | 1
Device failure (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 3
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cystitis klebsiella (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 2 | 0
Helicobacter infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 7
Pneumonia fungal (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 4
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 9
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 6 | 3
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 2
Nerve root injury (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Weight loss poor (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Akinesia (Nervous system disorders) | 2 | 3
Aphasia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Basilar artery thrombosis (Nervous system disorders) | 0 | 1
Bradykinesia (Nervous system disorders) | 2 | 3
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Cogwheel rigidity (Nervous system disorders) | 4 | 2
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3
Dysarthria (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 3
Epilepsy (Nervous system disorders) | 0 | 2
Freezing phenomenon (Nervous system disorders) | 2 | 1
Hypokinesia (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 2
Monoparesis (Nervous system disorders) | 0 | 1
On and off phenomenon (Nervous system disorders) | 3 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Parkinsonian gait (Nervous system disorders) | 3 | 2
Parkinsonian rest tremor (Nervous system disorders) | 3 | 2
Psychomotor hyperactivity (Nervous system disorders) | 2 | 0
Psychomotor skills impaired (Nervous system disorders) | 1 | 0
Quadriplegia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 5 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 4
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 3 | 6
Delirium (Psychiatric disorders) | 0 | 2
Delusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 4
Hallucination, visual (Psychiatric disorders) | 3 | 3
Insomnia (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Bladder trabeculation (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 3 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exelon Capsule (N=294) | Exelon Patch (N=288)
Constipation (Gastrointestinal disorders) | 21 | 21
Diarrhoea (Gastrointestinal disorders) | 27 | 14
Nausea (Gastrointestinal disorders) | 117 | 23
Vomiting (Gastrointestinal disorders) | 45 | 7
Application site erythema (General disorders) | 0 | 40
Fatigue (General disorders) | 19 | 13
Urinary tract infection (Infections and infestations) | 17 | 21
Fall (Injury, poisoning and procedural complications) | 48 | 49
Weight decreased (Investigations) | 19 | 18
Decreased appetite (Metabolism and nutrition disorders) | 18 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 16
Bradykinesia (Nervous system disorders) | 13 | 15
Dizziness (Nervous system disorders) | 26 | 21
Headache (Nervous system disorders) | 15 | 12
On and off phenomenon (Nervous system disorders) | 12 | 16
Parkinsonian gait (Nervous system disorders) | 15 | 12
Parkinsonian rest tremor (Nervous system disorders) | 69 | 26
Somnolence (Nervous system disorders) | 23 | 18
Anxiety (Psychiatric disorders) | 17 | 22
Confusional state (Psychiatric disorders) | 21 | 21
Depression (Psychiatric disorders) | 6 | 22
Hallucination (Psychiatric disorders) | 19 | 21
Hallucination, visual (Psychiatric disorders) | 12 | 16
Insomnia (Psychiatric disorders) | 14 | 23
Hypertension (Vascular disorders) | 16 | 12
Hypotension (Vascular disorders) | 22 | 10
Orthostatic hypotension (Vascular disorders) | 18 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.